CLINICAL TRIAL: NCT04556552
Title: Non-Invasive Vagal Nerve Stimulation in Opioid Use Disorders
Acronym: nVNS in OUDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); City University of New York (Other); Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, James Douglas Bremner, Professor of Psychiatry, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00117320; UG3DA048502 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Substance-Related Disorders; Substance Use Disorders; Substance Abuse, Intravenous; Substance Withdrawal; Substance Abuse; Opioid-use Disorder; Opioid Use Disorder, Severe; Opioid Use
Keywords: opioid use disorder; vagus nerve; vagal nerve; neuromodulation; vagus nerve stimulation; OUD
MeSH Terms: conditions — Substance-Related Disorders; Substance Abuse, Intravenous; Opioid-Related Disorders | interventions — Oxygen; Oxygen-15; Water

STUDY DESIGN:
Intervention Model Description: nVNS versus sham stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sham stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active non-invasive Vagal nerve stimulation (VNS) (Experimental): Active non-invasive Vagal Nerve Stimulation (nVNS) with opioid cues.
  Interventions: Device: Non invasive VN stimulation (nVNS); Drug: Oxygen (15-O) Water
- Sham stimulation (Sham Comparator): Sham stimulation of vagus with opioid cues
  Interventions: Drug: Oxygen (15-O) Water; Device: Sham Stimulation

INTERVENTIONS:
Device: Non invasive VN stimulation (nVNS) — Stimulation of vagus nerve with active device. Participants will be administered nVNS using the electroCore GammaCore-S non-invasive VNS device. The intensity of the stimulus will be adjusted by the user, to the maximum tolerable level to ensure nVNS without causing excessive pain, the burst frequency to 5 kHz, and the envelope frequency to 25 Hz.
  The duration of delivery will be 2 minutes, and the beginning will coincide with initiation of acquisition of the HR-PET scan which will be 90 seconds in duration; following an additional 8 minutes, a second VNS delivery will be administered, in conjunction with which another scan will be obtained.
  Arms: Active non-invasive Vagal nerve stimulation (VNS)
Drug: Oxygen (15-O) Water — Injection of radiolabelled water. H2[15-O] is a radioactive material. Each patient will have eight H2[15-O] blood flow scans. For each O-15 water scan 20 mCi of H2[15O] will be injected as an intravenous bolus.
  Other Names: radiolabelled water
Device: Sham Stimulation — Sham stimulation of vagus during opioid cue exposure. Each subject in the "SHAM" group will undergo the action of administering the intervention, but the device will be programmed such that the stimulation will not activate the vagus nerve.
  Arms: Sham stimulation

SUMMARY:
Subjects in this study will be patients with opioid use disorders (OUDs) based on DSM-5 criteria recruited from the greater Atlanta metropolitan region. Recruitment will be from treatment programs in the greater Atlanta Metropolitan Region including the DeKalb Community Service Board residential, detoxification and other treatment programs which with over 30,000 patient visits per year represents the largest treatment program in one of two urban counties in greater Atlanta.

This trial involves a second phase after completing an exploratory study in 20 patients with OUDs to assess different timing parameters of nVNS effects on sympathetic measures and symptoms of craving, as well as modelling to verify and iteratively refine the methods for vagal nerve stimulation. The investigators in this trial will then apply nVNS comparing active (N=10) to sham (N=10) in OUD patients recently started on medication, looking at opioid craving, brain functional response with HR-PET, and cardiovascular and inflammatory biomarker responses to imagery-induced opioid drug craving.

DETAILED DESCRIPTION:
Subjects in this study will be patients with opioid use disorders (OUDs) based on DSM-5 criteria recruited from the greater Atlanta metropolitan region. The metropolitan Atlanta area has about 2,623,744 persons age 12 or older. According to the Substance Abuse and Mental Health Services Administration (SAMHSA), 109,777 (4.18%) have non-medical use of prescription pain relievers, and 48,302 are estimated to have an opioid use disorder. This DSMP describes the UG3 phase which will study patients with OUDs early in the course of treatment. The Go-No Go criteria listed below have to be met to proceed to the UH3. Recruitment will be from treatment programs in the greater Atlanta Metropolitan Region including the DeKalb Community Service Board residential, detoxification and other treatment programs which with over 30,000 patient visits per year represents the largest treatment program in one of two urban counties in greater Atlanta.

The first UG3 phase will involve an exploratory study in 20 patients with OUDs to assess different timing parameters of nVNS effects on sympathetic measures and symptoms of craving, as well as modelling to verify and iteratively refine our methods for vagal nerve stimulation. The investigators in this trial will then apply nVNS in a pilot study comparing active (N=10) to sham (N=10) in OUD patients recently started on medication, looking at opioid craving, brain functional response with HR-PET, and cardiovascular and inflammatory biomarker responses to imagery-induced opioid drug craving. Brain function will be measured with high resolution positron emission tomography (HR-PET), autonomic function with wearable sensing devices, and biomarkers will be measured in blood, with an assessment of a broad range of stress responsive sympathetic, hormonal and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Subjects aged 18 and over who meet criteria for OUDs based on the Structured Clinical Interview for DSM-5 (SCID) interview and are stable on medication treatment.

Exclusion Criteria:

1. Positive pregnancy test
2. Meningitis
3. Traumatic brain injury
4. Neurological disorder or organic mental disorder
5. History of loss of consciousness greater than one minute
6. Current pregnancy or breastfeeding for women
7. Current or lifetime history of schizophrenia, schizoaffective disorder, or bulimia, based on the SCID
8. A history of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness
9. Evidence of a major medical or neurological illness that is based on the clinical judgment of the study psychiatrist
10. Active implantable device (i.e. pacemaker)
11. Carotid atherosclerosis
12. Cervical vagotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Douglas Bremner, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman FN, Nawar A, Nye JA, Choi J, Lambert TP, Robinson M, Gazi AH, Abbaraju V, Tomic N, Harrison AB, Jaquemet N, Mermin-Bunnell K, Mesfin H, Gray TA, Welsh JW, Dunn KE, Bikson M, Vaccarino V, Shah AJ, Inan OT, Bremner JD. Transcutaneous Cervical Vagus Nerve Stimulation Modulates Prefrontal Cortex Activity During Opioid Withdrawal in Individuals With Opioid Use Disorder. Neuromodulation. 2025 Dec;28(8):1396-1407. doi: 10.1016/j.neurom.2025.04.012. Epub 2025 Jun 23. PMID 40548916
- [Derived] Gazi AH, Harrison AB, Lambert TP, Obideen M, Alavi P, Murrah N, Shallenberger L, Driggers EG, Ortega RA, Washington BP, Walton KM, Welsh JW, Vaccarino V, Shah AJ, Tang YL, Gupta R, Back SE, Inan OT, Bremner JD. Transcutaneous cervical vagus nerve stimulation reduces behavioral and physiological manifestations of withdrawal in patients with opioid use disorder: A double-blind, randomized, sham-controlled pilot study. Brain Stimul. 2022 Sep-Oct;15(5):1206-1214. doi: 10.1016/j.brs.2022.08.017. Epub 2022 Aug 27. PMID 36041704

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Non-invasive Vagal Nerve Stimulation (VNS): Active non-invasive Vagal Nerve Stimulation (nVNS) with opioid cues.
  Non invasive VN stimulation (nVNS): Stimulation of vagus nerve with active device.
  Participants will be administered nVNS using the electroCore GammaCore-S non-invasive VNS device. The intensity of the stimulus will be adjusted by the user, to the maximum tolerable level to ensure nVNS without causing excessive pain, the burst frequency to 5 kHz, and the envelope frequency to 25 Hz.
  The duration of delivery will be 2 minutes, and the beginning will coincide with initiation of acquisition of the HR-PET scan which will be 90 seconds in duration; following an additional 8 minutes, a second VNS delivery will be administered, in conjunction with which another scan will be obtained.
  Oxygen (15-O) Water: Injection of radiolabelled water. H2[15-O] is a radioactive material. Each patient will have eight H2[15-O] blood flow scans. For each O-15 water scan 20 mCi of H2[15O] will be injected as an intravenous bolus.
Period: Overall Study
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Started | 12 | 8
Completed | 11 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Claustrophobia | 0 | 1
Not completed — Inability to continue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.857) | 48.375 (9.366) | 44.25 (15.348)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 7 | 19
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 3 | 5 | 8
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Opioid Craving Using Visual Analogue Scale
Description: Opioid craving will be measured based on Visual Analogue Scale (VAS) VAS consist in 10-point lines anchored with "not at all" on one end and "extremely" on the other where participants report the extent to which they felt any craving for opiates, severity of withdrawal symptoms, and the extent to which the study intervention has helped to ease the cravings. Total possible score ranges from 0 to100, with 100 correlating with worse study outcome.
Time Frame: Baseline, 5 minutes post-intervention
Population: Number analyzed in one or more rows differs from overall number analyzed because some data was not collected for technical reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 11 | 7
score on a scale
  Baseline | 3.909 (3.048) | 6 (2.160)
  5 min post-intervention: number analyzed (Participants) | 11 | 6
  5 min post-intervention | 4.556 (2.186) | 5.5 (3.937)

2. Primary Outcome: Heart Rate (HR)
Description: Heart rate will be measured after cue. Decreased HR correlates with better outcome.
Time Frame: Baseline, two minutes post-intervention
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 11 | 6
bpm
  Baseline | 64.357 (8.275) | 61.575 (10.715)
  Two minutes post-intervention | 64.192 (9.960) | 59.003 (10.182)

3. Primary Outcome: Pre-ejection Period (PEP)
Description: Pre-ejection Period (PEP) is a marker of cardiac sympathetic tone that is increased with blocked sympathetic function. Higher PEP correlates with better outcome.
Time Frame: Baseline, 2 minutes post-intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 11 | 6
seconds
  Baseline | 0.048 (0.033) | 0.069 (0.035)
  2 minutes post-intervention | 0.050 (0.0320) | 0.066 (0.0312)

4. Primary Outcome: Photoplethysmography (PPG) Amplitude
Description: Photoplethysmography (PPG) amplitude reflects vasoconstriction in figure blood vessel. PPG amplitude is increased with blocked sympathetic tone and higher PPG correlates with better outcome.
Time Frame: Baseline, 2 minutes post-intervention
Measure: Mean (Standard Deviation); unit: AU (arbitrary units)
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 11 | 6
AU (arbitrary units)
  Baseline | 1.411 (1.285) | 1.684 (0.838)
  2 minutes post-intervention | 1.162 (2.312) | 1.459 (0.873)

5. Primary Outcome: Brain Blood Flow in the Anterior Cingulate With VNS Paired With Opioid Use Videos
Description: Brain blood flow measured with Positron Emission Tomography (PET) and radiolabeled water at baseline and 2 min post-intervention during viewing of neutral videos and with active and Sham VNS stimulation paired with opioid use videos. Brain blood flow was measured in mL per 100 g of tissue per minute (mL/100g/min) normalized to a reference of 50 ml/100 g of tissue per minute.
Time Frame: Baseline, 2 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mL/100g/min
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 7 | 4
mL/100g/min
  Baseline | 56.1 (40.7) | 44.5 (18.1)
  2 minutes post-intervention | 40.2 (10.2) | 29.2 (12.2)

6. Secondary Outcome: Levels of Interleukin 6 (IL-6)
Description: IL-6 is an inflammatory marker. Reduced levels of IL-6 correlate with better outcome.
Time Frame: Baseline, 2 minutes post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
Number analyzed (Participants) | 10 | 5
pg/ml
  Baseline | 1.4 (0.8) | 4.0 (3.1)
  2 min post-intervention: number analyzed (Participants) | 7 | 4
  2 min post-intervention | 2.6 (2.6) | 3.9 (3.1)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 5 min.
Arm/Group | Active Non-invasive Vagal Nerve Stimulation (VNS) | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04556552/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04556552/ICF_000.pdf